CLINICAL TRIAL: NCT06351917
Title: Effect of Topical PlexoZome® Levagen® Spray on Relief of Post Exercise Knee Joint Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEVEXE
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-04

CONDITIONS: Knee Joint Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PlexoZome® Levagen® (Experimental): PlexoZome® Levagen® topical spray solution applied as 3 full pumps on the affected knee area providing 5.6mg of active per 3 pumps.
  Interventions: Drug: PlexoZome® Levagen® topical spray solution
- Placebo Comparator (Placebo Comparator): Placebo topical spray solution applied as 3 full pumps on the affected knee area providing 0mg of active per 3 pumps.
  Interventions: Drug: Placebo topical spray solution

INTERVENTIONS:
Drug: PlexoZome® Levagen® topical spray solution — PlexoZome® Levagen® topical spray solution 10mg/g providing 1.8mg active per pump
  Arms: PlexoZome® Levagen®
Drug: Placebo topical spray solution — Placebo topical spray solution topical spray solution 0mg/g providing 0mg active per pump
  Arms: Placebo Comparator

SUMMARY:
This is a randomised, double-blind, placebo controlled, 2 arm parallel clinical trial to evaluate the effect of topical PlexoZome® Levagen® spray on relief of post exercise knee joint pain in healthy adults compared to placebo over 4 weeks duration.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years
* Generally healthy
* Able to provide informed consent
* Undertaking regular exercise
* Experiencing post exercise knee pain of at least 3 (on a 0-10 scale) at least 2 times in previous 4 weeks
* Agree not to change current diet and/or exercise frequency or intensity

Exclusion Criteria:

* Serious illness( 1 ) e.g., mood disorders such as depression, anxiety or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Unstable illness( 2 ) e.g., diabetes and thyroid gland dysfunction
* Current malignancy (excluding BCC) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy
* Active smokers, nicotine use, alcohol( 3 ) or drug (prescription or illegal substances) abuse
* Allergic to any of the ingredients in the active or placebo formula
* Pregnant or lactating women
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion

Footnotes

( 1 )A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

( 2 )An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity.

( 3 )Chronic past and/or current alcohol use (>14 alcohol drinks/week)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Joint pain | Up to 5 knee pain treatment events for up to 4 weeks
  Joint pain via Visual Analogue Scale (VAS) Pain Scale which requires a pain rating from 1 to 10 with 1 indicating no pain and 10 indicating worse pain possible.

SECONDARY OUTCOMES:
Time to pain relief | Up to 5 knee pain treatment events for up to 4 weeks
  Time to pain relief via Visual Analogue Scale (VAS) Pain Scale which requires a pain rating from 1 to 10 with 1 indicating no pain and 10 indicating worse pain possible.
Number of Adverse Events | Enrolment period
  Number of Adverse Events via AE monitoring
Severity of Adverse Events | Enrolment period
  Severity of Adverse Events via AE monitoring
Rescue medication use | Up to 5 knee pain treatment events for up to 4 weeks
  Rescue medication use via self-report

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia